CLINICAL TRIAL: NCT03246542
Title: Association Between the Quantitative Assessment of Schistocytes in Peripheral Blood Smear and Prognosis of Patient Initially Diagnosed as HELLP Syndrome.
Brief Title: Promising Bimarker Prediction of Outcome of HELLP Syndrome.
Status: Completed | Type: Observational
Sponsor: AYMAN ABDELKADER MOHAMED ABDELKADER (Other)
Responsible Party: Sponsor-Investigator, AYMAN ABDELKADER MOHAMED ABDELKADER, doctor, Ain Shams Maternity Hospital
Organization: Ain Shams Maternity Hospital (Other)
Other Study IDs: AAMABDELKADER 4
Record Dates: First submitted 2017-07-23; First posted 2017-08-11 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Pre-Eclampsia, Severe; HELLP Syndrome; Microangiopathy
MeSH Terms: conditions — Pre-Eclampsia; HELLP Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: shistocytes percentage

SUMMARY:
HELLP syndrome is a life-threatening obstetric complication usually considered to be a variant or complication of pre-eclampsia. And may occasionally be confused with other diseases complicating pregnancy such as acute fatty liver of pregnancy, gastroenteritis, hepatitis, appendicitis, gallbladder disease, immune thrombocytopenia, lupus flare, antiphospholipid syndrome, hemolytic-uremic syndrome, thrombotic thrombocytopenic purpura, and nonalcoholic fatty liver disease. The distinction between thrombotic thrombocytopenic purpura-hemolytic uremic syndrome and severe preeclampsia is important for therapeutic and prognostic reasons. However, the clinical and histological features are so similar that establishing the correct diagnosis is often difficult; furthermore, these disorders may occur concurrently.

DETAILED DESCRIPTION:
When TTP/HUS does occur during pregnancy, they often are confused initially with obstetric diagnoses such as severe preeclampsia; hemolysis, elevated liver enzymes and low platelets (HELLP) syndrome; acute fatty liver of pregnancy; eclampsia, and antiphospholipid antibody syndrome. This might be related to the fact that the disease entity is rare and often is unexpected. Nevertheless, a delay in diagnosis of TTP/HUS may result in life-threatening maternal and fetal consequences. Aim of the current study was to compare the quantitative assessment of schistocytes in peripheral blood smear between women initially diagnosed as HELLP syndrome who showed no spontaneous resolution within 48 hrs after delivery and those who showed spontaneous resolution within 48 hrs after delivery which may help in decreasing the maternal mortality rate .

ELIGIBILITY:
Inclusion Criteria:

* Gestational age more than 20 weeks.
* Age from18 to 40 years old.
* Fulfilled criteria for the diagnosis of severe preeclampsia.
* Fulfilled criteria for the diagnosis of HELLP syndrome.

Diagnostic criteria for severe preeclampsia(one of the following):

* Blood pressure of 160 mm Hg systolic or higher or 110 mm Hg diastolic or higher on two occasions at least 6 hours apart while the patient is on bed rest (unless antihypertensive therapy is intiated befor this time).
* New onest Cerebral or visual disturbances.
* Pulmonary edema or cyanosis.
* Sever persistant epigastric or right upper-quadrant pain unresponsive to medication and not accounted for by alternative diagnosis, or both.
* Impaired liver function as indicated by abnormally elevated blood concentration of liver enzymes (to twic normal concentration).
* Thrombocytopenia (platlet count less than 100, 000 per microliter.

Diagnostic criteria for HELLP syndrome:

* Hemolysis documented by an increased LDH level and progressive anemia .
* Hepatic dysfunction documented by an LDH level >600 IU/L, elevated liver enzymes documented by AST >40 IU/L, ALT>40 IU/L, or both .
* Thrombocytopenia documented by a platelet nadir less than 150, 000 cells/mm³. Thrombocytopenia is subclassified as class one HELLP syndrome: platelet nadir ≤50, 000 cells/mm³, class two HELLP syndrome: platelet nadir ≤100, 000 cells/mm³, or class three HELLP syndrome: platelet nadir ≤150, 000 cells/mm³..

Anticepation of Microangiopathic Hemolytic Anemia:

Thrombotic thrombocytopenic purpura-hemolytic uremic syndrome should be considered in all pregnant women with severe thrombocytopenia, severe anemia, and elevated lactate dehydrogenase enzyme.

Exclusion Criteria: any non included criteria

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 100 women with an initial diagnosis of HELLP syndrome were recruited in the study.
  Blood sample taken within 12hrs peripartum and patients followed up 48hrs after delivery and subdivided in to 2 groups according to improvement or deterioration after 48hrs after delivery .
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
laboratory changes after 48 hours of delivery | 48 hours
  full blood count, liver function tests( AST, ALT, Bilirubin), kidney function (serum creatinine level), coagulation profile (INR, PTT, PT)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2014-09-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT03246542/Prot_000.pdf
  • Statistical Analysis Plan (2016-01-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT03246542/SAP_001.pdf